CLINICAL TRIAL: NCT02981381
Title: Synchronized TMS for Posttraumatic Stress Disorder and Comorbid Depressive Symptoms
Brief Title: Synchronized Transcranial Magnetic Stimulation for PTSD
Acronym: sTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence VA Medical Center (U.S. Federal Agency)
Collaborators: Wave Neuroscience (Industry)
Responsible Party: Principal Investigator, Noah S. Philip, MD, Psychiatrist, Providence VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-004; 1010584-1 (Other: Veteran's IRB of Northern New England (VINNE))
Record Dates: First submitted 2016-10-24; First posted 2016-12-05 (Estimated); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: PTSD; Depression
Keywords: sTMS; NeoSync; NEST; synchronous; non-invasive neuromodulation; TMS; Transcranial Magnetic Stimulation; PTSD; EEG; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active sTMS (NEST-1) (Experimental): Subjects randomized to this group will receive 20 active synchronized Transcranial Magnetic Stimulation (sTMS) treatments (30 minutes each) over a period of 40 calendar days. Treatment windows will be 10 calendar days to complete 5 active sTMS sessions. Serial assessments will be completed every 5 sessions. Post-treatment (PT1) endpoint assessments will take place on the last day of active sTMS.
  Participants that elect to participate in the open-label continuation phase, will receive an additional 20 sTMS treatments (using the NEST-2 device), following the same administration structure as the sham-control series.
  Participants will return to complete post-treatment follow-up assessments (PT2) 1 month after their last treatment session (either PT1 or OL PT1).
  Interventions: Device: NEST-1; Device: NEST-2
- Sham sTMS (SHAM) (Sham Comparator): Subjects randomized to this group will receive 20 sham synchronized Transcranial Magnetic Stimulation (sTMS) treatments (30 minutes each) over a period of 40 calendar days. Treatment windows will be 10 calendar days to complete 5 sham sessions. Serial assessments will be completed every 5 sessions. Post-treatment (PT1) endpoint assessments will take place immediately after the final sham session.
  Participants that elect to participate in the open-label continuation phase, will receive 20 sTMS treatments (using the NEST-2 device), following the same administration structure as the sham-control series.
  Participants will return to complete post-treatment follow-up assessments (PT2) 1 month after their last treatment session (either PT1 or OL PT1).
  Interventions: Device: SHAM; Device: NEST-2

INTERVENTIONS:
Device: NEST-1 — The NeoSync EEG Synchronized TMS (NEST) is an electromechanical medical device that produces and delivers a sinusoidal magnetic field to areas of the brain in the treatment of PTSD. The device includes an EEG recording module that is used to record individualized alpha frequency (IAF) on randomized personal passport modules (PPM) pre-assigned to be NEST-1 compatible.
  Other Names: Active sTMS; NeoSync EEG Synchronized TMS
  Arms: Active sTMS (NEST-1)
Device: SHAM — The SHAM NeoSync EEG Synchronized TMS (NEST) is a device, identical to the active NEST-1 device, that is configured to simulate the delivery of active treatment without actively delivering sTMS therapy. The device includes an EEG recording module that is used to record individualized alpha frequency (IAF) on randomized personal passport modules (PPM) pre-assigned to be SHAM compatible.
  Other Names: NEST-1 Sham Comparator
  Arms: Sham sTMS (SHAM)
Device: NEST-2 — The open-label NeoSync EEG Synchronized TMS (NEST) that produces and delivers a sinusoidal magnetic field to areas of the brain in the treatment of PTSD. The device is distinct in both color and sound both SHAM and NEST-1 devices. PPMs corresponding with both SHAM and NEST-1 devices are compatible with the NEST-2 device.
  Other Names: Open-label sTMS; NeoSync EEG Synchronized TMS

SUMMARY:
The investigators propose a small, two-site, sham-controlled pilot study of synchronized Transcranial Magnetic Stimulation (sTMS) in patients with comorbid post-traumatic stress disorder (PTSD) and depression. It is hypothesized that sTMS will be effective for PTSD and mood symptoms.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a highly prevalent psychiatric disorder associated with high degrees of comorbidity (e.g., major depressive disorder), poor quality of life, and significant social and occupational dysfunction. Currently available evidence-based pharmacological and psychological treatments for PTSD have only modest efficacy, and thus further research is necessary to develop treatment approaches in order to ameliorate the current disparity between disorder impact and prevalence, and effective therapies.

The use of non-invasive neuromodulation techniques, such as repetitive transcranial magnetic stimulation (rTMS), in an outpatient setting, has shown to be effective in reducing symptoms in various mental disorders, including PTSD and major depressive disorder (MDD). Research examining the use of rTMS for PTSD still remain limited, the majority of findings pertain to rTMS in MDD cohorts, which excluded individuals with PTSD. Given the high rate of PTSD with MDD comorbidity, additional studies examining this comorbid population are necessary.

Furthermore, rTMS treatment parameters and duration are rather time consuming for patients, requiring that patient travel to an outpatient facility daily, for 6 to 8 weeks, for 30 to 40 minutes each day. This can be an inconvenience and poses an additional burden for individuals that already struggle with societal integration and social/occupational dysfunction. Thus, further exploration and development of non-invasive brain stimulatory devices with the same (or better) effectiveness as rTMS, that can be adapted to be utilized in an at home setting, would revolutionize the treatment of PTSD.

The synchronized transcranial magnetic stimulation (sTMS, NeoSync Inc.) device provides the possibility of the fore mentioned therapeutic development. The sTMS device employs 3 transversely rotating, to deliver low energy, sinusoidal magnetic fields synchronized to an individuals' intrinsic alpha frequency (IAF). Preliminary data has shown that sTMS can effectively reduce depressive symptoms in MDD. Additionally, the investigators' preliminary examination of IAF in participants with comorbid PTSD and depressive symptoms, has illuminated the feasibility of this modality as a treatment approach for PTSD comorbid with MDD.

This study is a prospective, sham-controlled, trial of sTMS delivered to patients who are symptomatic despite ongoing pharmacotherapy for PTSD and mood symptoms. Eligible subjects will be randomized using to receive 4 weeks (5 daily sessions per week) of either sham or active sTMS treatment. Clinical and self-report assessments will be completed at baseline, sham/control series endpoint, and 1 month after the final treatment session. An optional open-label continuation phase will be offered to all study participants who complete the sham-control phase of this study, and additional endpoint assessments will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Veteran;
* MRI safe;
* Meet Diagnostic and Statistical Manual, Fifth Edition (DSM 5) criterion for PTSD (acute or chronic, confirmed by the Clinician Administered PTSD Scale (CAPS) and at least moderate severity defined by a PCL-5 score > 33); AND at least moderate depressive symptom severity (defined by QIDS-SR score > or equal to 11) at baseline visit. Individuals with bipolar II or otherwise unspecified who are currently in a depressed episode are eligible;
* Baseline score of "moderately ill" or worse on the Clinical Global Impressions-Severity (CGI-S);
* Stable psychotropic regimen for at least 6 weeks prior to baseline and willing to maintain current dose and regimen throughout study, or no psychotropic medication at all;
* If female and of child bearing potential, must agree to use an acceptable method of birth control for the duration of the study treatment period;
* Be willing and able to comply with all study related procedures and visits;
* Be capable of independently reading and understanding all patient information materials and giving written informed consent.

Exclusion Criteria:

* Pregnant or lactating, or planning on becoming pregnant within the next 3 months;
* Lifetime history of loss of consciousness (>10 minutes) due to head injury, or lifetime history of head injury with documented evidence of brain injury;
* Current (or past) significant neurological disorders (seizure disorder, primary or secondary central nervous system (CNS) tumors, stroke, cerebral aneurysm);
* Unstable medical illness, or significant absence of appropriate medical care;
* Current axis I primary psychotic disorder or Bipolar I disorder;
* Active (within the last month) moderate or severe substance (excluding nicotine/caffeine) abuse disorders. Individuals on stable (>3 months), monitored opiate agonist therapy may be included at investigator's discretion;
* Past failed treatment with rTMS or electroconvulsive therapy (ECT); any past treatment with deep brain stimulation or vagus nerve stimulation;
* Have an active suicidal intent or plan, or in the opinion of the investigator, is likely to attempt suicide in the next 6 months;
* Presence of condition or circumstance with potential to prevent study completion;
* Inability to obtain sufficient EEG to calibrate study device.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah S Philip, MD, Principal Investigator — Study Principal Investigator
Locations (2):
- United States (2):
  - Providence VAMC, Providence, Rhode Island
  - White River Junction VAMC, White River Junction, Vermont

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active sTMS (NEST-1): Subjects randomized to this group will receive 20 active synchronized Transcranial Magnetic Stimulation (sTMS) treatments (30 minutes each) over a period of 40 calendar days. Treatment windows will be 10 calendar days to complete 5 active sTMS sessions. Serial assessments will be completed every 5 sessions. Post-treatment (PT1) endpoint assessments will take place on the last day of active sTMS.
  Participants that elect to participate in the open-label continuation phase, will receive an additional 20 sTMS treatments (using the NEST-2 device), following the same administration structure as the sham-control series.
  Participants will return to complete post-treatment follow-up assessments (PT2) 1 month after their last treatment session (either PT1 or OL PT1).
  NEST-1: The NeoSync EEG Synchronized TMS (NEST) is an electromechanical medical device that produces and delivers a sinusoidal magnetic field to areas of the brain in the treatment of PTSD. The device includes an EEG recording module that is used to record individualized alpha frequency (IAF) on randomized personal passport modules (PPM) pre-assigned to be NEST-1 compatible.
  NEST-2: The open-label NeoSync EEG Synchronized TMS (NEST) that produces and delivers a sinusoidal magnetic field to areas of the brain in the treatment of PTSD. The device is distinct in both color and sound both SHAM and NEST-1 devices. PPMs corresponding with both SHAM and NEST-1 devices are compatible with the NEST-2 device.
- Sham sTMS (SHAM): Subjects randomized to this group will receive 20 sham synchronized Transcranial Magnetic Stimulation (sTMS) treatments (30 minutes each) over a period of 40 calendar days. Treatment windows will be 10 calendar days to complete 5 sham sessions. Serial assessments will be completed every 5 sessions. Post-treatment (PT1) endpoint assessments will take place immediately after the final sham session.
  Participants that elect to participate in the open-label continuation phase, will receive 20 sTMS treatments (using the NEST-2 device), following the same administration structure as the sham-control series.
  Participants will return to complete post-treatment follow-up assessments (PT2) 1 month after their last treatment session (either PT1 or OL PT1).
  SHAM: The SHAM NeoSync EEG Synchronized TMS (NEST) is a device, identical to the active NEST-1 device, that is configured to simulate the delivery of active treatment without actively delivering sTMS therapy. The device includes an EEG recording module that is used to record individualized alpha frequency (IAF) on randomized personal passport modules (PPM) pre-assigned to be SHAM compatible.
  NEST-2: The open-label NeoSync EEG Synchronized TMS (NEST) that produces and delivers a sinusoidal magnetic field to areas of the brain in the treatment of PTSD. The device is distinct in both color and sound both SHAM and NEST-1 devices. PPMs corresponding with both SHAM and NEST-1 devices are compatible with the NEST-2 device.
Period: Double Blind Phase
Arm/Group | Active sTMS (NEST-1) | Sham sTMS (SHAM)
Started | 10 | 13
Completed | 7 | 12
Not Completed | 3 | 1
Period: Optional Unblinded sTMS
Arm/Group | Active sTMS (NEST-1) | Sham sTMS (SHAM)
Started | 5 | 12
Completed | 5 | 10
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active sTMS (NEST-1) | Sham sTMS (SHAM) | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 13 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 9 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 11 | 19
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: PCL-5 Total Score Change
Description: The PTSD checklist (PCL-5) will be used to assess PTSD symptom severity pre- and post-treatment. The change in total PCL-5 score from Baseline (Day 0) to endpoint (PT1) compared between active treatment and sham-controlled groups. If a participant does not complete PT1, last observation carried forward (LOCF) will be used. A 50% reduction in scores from Baseline scores to PT1 indicates clinical response to treatment (active sTMS vs. sham), and remission is defined by a post-treatment score below the threshold score published for the PCL-5.
  The PCL-5 (PTSD Checklist for DSM-5) is a 20-item self-report measure used to assess the presence and severity of posttraumatic stress disorder (PTSD) symptoms; scores go from 0 to 80, where higher scores indicate greater severity. A score greater than 33 is typically used to indicate severity sufficient for a PTSD diagnosis. Items are rated from 0 (Not at all) to 4 (extremely) bothersome.
Time Frame: 1 month after final treatment (approximately 70 days total)
Measure: Mean (Standard Deviation); unit: Units on a scale (PCL-5)
Arm/Group | Active sTMS (NEST-1) | Sham sTMS (SHAM)
Number analyzed (Participants) | 10 | 13
Units on a scale (PCL-5) | 50.1 (7.4) | 49.2 (9.3)

ADVERSE EVENTS:
Time Frame: 1 month after final treatment (approximately 70 days total).
Description: Adverse event reporting indicates all events in the groups examined (i.e., include both double-blind and unblinded study periods). Reported adverse events include those observed during the open-label period (i.e., all reported adverse events occurred during the double-blind phase of the study).
Arm/Group | Active sTMS (NEST-1) | Sham sTMS (SHAM)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/12
Other Adverse Events (participants affected / at risk) | 0/7 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT02981381/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT02981381/ICF_001.pdf